CLINICAL TRIAL: NCT03573830
Title: Randomized Control Trial of an Intervention to Increase Perceived Safety Benefit of Booster Seats Among Parents of Children 4 to 8 Years Old in Canada.
Brief Title: Randomized Control Trial of Booster Seat Education Material to Increase Perceived Benefit Among Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Child and Family Research Institute (Other)
Responsible Party: Principal Investigator, Mariana Brussoni, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H14-01569
Record Dates: First submitted 2018-06-05; First posted 2018-06-29 (Actual); Results first posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Wounds and Injuries
Keywords: Child Passenger Injury; Child Restraint Systems; Traffic Accidents
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: PARTICIPANT MASKING: Participants will be told the purpose of the study is to evaluate parents' reactions to two different information materials about booster seats and seatbelts.
  INVESTIGATOR MASKING: The study will be conducted entirely online using a online research platform, so allocation will be masked to all investigators.
  OUTCOMES ASSESSOR MASKING: Outcome evaluation will be conducted online using an online survey tool, so allocation will be masked to outcome assessors.
  STATISTICAL ANALYSIS: Allocation in the online survey will be coded using random numbers unknown to the person conducting statistical analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Current material (Active Comparator): Participants in this arm will be shown the online Transport Canada Material that is currently available at: https://www.tc.gc.ca/en/services/road/child-car-seat-safety/installing-using-child-car-seat-booster-seat-seat-belt/stage-3-booster-seats.html
  Interventions: Behavioral: Transport Canada material
- Enhanced material (Experimental): Participants in this arm will be shown an enhanced version of the online Transport Canada Material, which includes an introduction explaining how booster seats prevent injuries caused by seat belts.
  Interventions: Behavioral: Enhanced material

INTERVENTIONS:
Behavioral: Transport Canada material — The current Transport Canada booster seat education material focuses on imparting guidelines; that is, it describes, in plain language, the minimum and maximum ages, heights, and weights to determine when a child should use a booster seat, and when it is safe for a child to use only the seat belt. This material does not describe the principle of operation of seat belts (i.e., redirecting crash forces to the rib cage and pelvis), nor the principle of operation of booster seats (i.e., ensuring the seat belt is placed correctly across the chest and hips).
  Other Names: Current Transport Canada material
  Arms: Current material
Behavioral: Enhanced material — Enhancements to the booster seat education material were developed based on the hypothesis that parents would better appreciate the additional injury risk reduction afforded by booster seats, if they understand that: (1) seat belts prevent injuries by redirecting crash forces to stronger parts of the body (i.e., rib cage and pelvis); and (2), without booster seats, children would wear the seat belt on their abdomen and neck, which directs crash forces to more vulnerable anatomical structures (i.e., internal organs and spine).
  Other Names: Enhanced Transport Canada material
  Arms: Enhanced material

SUMMARY:
Seat belts protect people from injuries by diverting crash forces to stronger anatomical structures: the rib cage and the pelvis. Children between the ages of 4 and 8 years are typically not tall enough to wear the seat belt correctly across the chest and hips, and instead wear it on their abdomen and neck. When worn in this way, seat belts direct crash forces to these parts of the body, potentially causing serious damage to internal organs and the spine. For this reason, children of these ages need to use a booster seat; a safety device that prevents seat belt related injuries by raising the child and ensuring the straps are correctly worn across the thorax and hips. In Canada, half of the children who should be using booster seats are prematurely restrained using only the seat belt. The present research project seeks to develop and test a novel intervention to encourage booster seat use.

Many Canadian provinces have enacted laws mandating use, and have developed and implemented evidence-based education programs. Despite these efforts, new approaches to encourage booster seat use are required. In 2010, more than 10 years after booster seats became mandatory, the rate of utilization in the Canadian provinces of Ontario and Quebec was still low (25%). Furthermore, recent research indicates that parents' perception of the safety benefit of booster seats is the strongest predictor of use, yet no study to date has tested an education intervention that increases perceived benefit; instead, these interventions focus on teaching guidelines (i.e., minimum and maximum age, height, and weight to determine when a child should use a booster seat, and when it is safe for a child to use only the seat belt).

The present approach to encouraging booster seat use is novel, because it increases perceived benefit by teaching two principles: (1) seat belts prevent injuries by redirecting crash forces to stronger parts of the body (rib cage and pelvis); and (2), without booster seats, children would wear the seat belt on their abdomen and neck, which directs crash forces to more vulnerable anatomical structures (internal organs and spine). Once parents grasp these two principles, they are expected to better appreciate the safety benefit of booster seats and, thus, be more likely to use them.

DETAILED DESCRIPTION:
The education material currently available in the Transport Canada website will be enhanced, by adding an introduction that describes how seat belts and booster seats work (i.e., these devices help redirect crash forces to stronger parts to the body: rib cage and pelvis).

Objective of the trial: To determine if the enhanced material is better than the current Transport Canada information at increasing perceived safety benefit and intention to use booster seats.

Design: Concurrent two-group parallel randomized controlled trial.

Randomization: Block randomization will be used to assign participants to either intervention or control groups. Participants and researchers will be blinded to allocation.

Participants. 303 mothers and 303 fathers of children 4 to 8 years old will be invited to participate, irrespective of whether they use booster seats always, occasionally, or never. A sample of 606 participants provides sufficient power to detect a mean difference in perceived benefit that separates those parents who consistently restrain their child in booster seats from those who do not. Sample size was estimated with the TwoSampleMean function for trials that test superiority of interventions (TrialSize package for R). Participants in the trial will receive $1/each for the completion of the survey. Based on information from studies with similar characteristics, the expected response rate is 40%.

Setting and Procedures. The trial will be conducted entirely online. Participants will be recruited through an online market research firm, Maru/Matchbox, which maintains a nationwide panel of 130,000 individuals whose distribution represents the Canadian population. Maru/Matchbox will send an email invitation to participate along with a link to the online survey. The landing page of the survey will provide description of the study for parents to read. The online survey will be set up in such a way that participants won't be able to start answering questions, unless they consent by clicking the "I agree" button. Participants, will be advised to print and keep a copy of the consent form either as PDF or as hard copy. After consenting to participate, the online trial will proceed as follows:

1. Participants will complete a baseline questionnaire.
2. The system will randomly assign the participant to either the intervention or the control group. Randomization will be stratified by sex, child age, and jurisdiction to ensure both groups are equal.
3. Participants in the intervention group will be presented the enhanced booster seat material, while participants in the control group will be presented the current Transport Canada booster seat material. Material provided to both groups will be stripped of logos (Transport Canada logos and corporate identity), but will be properly cited.
4. Participants will complete post-intervention questionnaire.
5. Participants in the intervention group will be asked one or two questions to ensure they did not misunderstood the information in an unintended way. If a parent answers incorrectly, the system will clarify the information immediately after.
6. Participants in the control group will be given the option to view the enhanced booster seat material, in order to give them the opportunity to benefit from the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children 4 thorough 8 years old
* Residing in any Canadian Province
* Fluent in English
* Drive with their child at least once a month

Exclusion Criteria:

- Child has a physical condition that requires special transportation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 731 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2018-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Brussoni, PhD, Principal Investigator — University of British Columbia, BC Children's Hospital Research Institute
Locations (1):
- British Columbia Children's Hospital Research Institute, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
The data set and supporting documents will be available from Dr. Brussoni upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: until 2025
Access Criteria: Amy scholarly requests will be considered.

REFERENCES:
- [Background] Cunningham CE, Bruce BS, Snowdon AW, Chen Y, Kolga C, Piotrowski C, Warda L, Correale H, Clark E, Barwick M. Modeling improvements in booster seat use: a discrete choice conjoint experiment. Accid Anal Prev. 2011 Nov;43(6):1999-2009. doi: 10.1016/j.aap.2011.05.018. Epub 2011 Jun 25. PMID 21819828
- [Background] Committee on Injury, Violence, and Poison Prevention; Durbin DR. Child passenger safety. Pediatrics. 2011 Apr;127(4):788-93. doi: 10.1542/peds.2011-0213. Epub 2011 Mar 21. PMID 21422088
- [Background] Ishikawa T, Jiang A, Brussoni M, Reyna V, Weldon B, Bruce B, Pike I. Perceptions of injury risk associated with booster seats and seatbelts: the ejection stereotype hypothesis. Hypothesis Journal 15(1): e1.
- [Background] A. W. Snowdon, A. Hussein, E. Ahmed, "Canadian National Survey on Child Restraint Use 2010" (AUTO21, 2011). https://www.tc.gc.ca/eng/motorvehiclesafety/resources-researchstats-child-restraint-survey-2010-1207.htm
- See also: Transport Canada information on booster seats — https://tc.canada.ca/en/road-transportation/child-car-seat-safety/stage-3-booster-seats

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited online, between the 10th and the 27th of December 2018, through a market research service, Maru Blue, which keeps a database of 130,000 individuals who have consented to receive invitations to online surveys. Individuals registered in the database were sent an email invitation, which included a link to our online survey.
Pre-assignment Details: Our target sample size was 606, as stated in the protocol. However, we were able to enroll more than our target: 731
Groups:
- Current Material: Participants in this arm were shown the online Transport Canada Material that is was available at the time: https://tc.canada.ca/en/road-transportation/child-car-seat-safety/stage-3-booster-seats
  Transport Canada material: The current Transport Canada booster seat education material focuses on imparting guidelines; that is, it describes, in plain language, the minimum and maximum ages, heights, and weights to determine when a child should use a booster seat, and when it is safe for a child to use only the seat belt. This material does not describe the principle of operation of seat belts (i.e., redirecting crash forces to the rib cage and pelvis), nor the principle of operation of booster seats (i.e., ensuring the seat belt is placed correctly across the chest and hips).
- Enhanced Material: Participants in this arm were shown an enhanced version of the online Transport Canada Material, which includes an introduction explaining how booster seats prevent injuries caused by seat belts.
  Enhanced material: Enhancements to the booster seat education material were developed based on the hypothesis that parents would better appreciate the additional injury risk reduction afforded by booster seats, if they understand that: (1) seat belts prevent injuries by redirecting crash forces to stronger parts of the body (i.e., rib cage and pelvis); and (2), without booster seats, children would wear the seat belt on their abdomen and neck, which directs crash forces to more vulnerable anatomical structures (i.e., internal organs and spine).
Period: Overall Study
Arm/Group | Current Material | Enhanced Material
Started | 364 | 367
Reviewed Assigned Material (Whether participants completed their assigned intervention.) | 364 (All participants assigned to this arm reviewed their assigned material.) | 360 (360 reviewed their assigned material:Transport Canada information plus the enhanced material.)
Completed | 360 | 360
Not Completed | 4 | 7
Not completed — Dropped without completing treatment | 0 | 7
Not completed — Lost to Follow-up | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Current Material | Enhanced Material | Total
Number analyzed (Participants) | 364 | 367 | 731
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.40 (6.98) | 39.16 (7.10) | 38.78 (7.04)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Mothers | 191 | 199 | 390
  Fathers | 173 | 168 | 341
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Education [Count of Participants; unit: Participants]
  No certificate, diploma or degree | 14 | 18 | 32
  High school certificate or equivalent | 40 | 36 | 76
  Apprenticeship or trades | 55 | 52 | 107
  University certificate or diploma | 38 | 38 | 76
  College, CEGEP or equivalent | 84 | 68 | 152
  Bachelor's degree | 62 | 89 | 151
  Master's degree | 59 | 54 | 113
  PhD, MD, Dentist, or equivalent | 12 | 12 | 24
Number of children [Count of Participants; unit: Participants]
  One child | 74 | 81 | 155
  Two children | 186 | 166 | 352
  Three children | 62 | 83 | 145
  Four or more | 42 | 37 | 79
Language spoken at home [Count of Participants; unit: Participants]
  English | 343 | 339 | 682
  Other language | 21 | 28 | 49
Perceived Benefit of Booster Seats [Mean (Standard Deviation); unit: Scores on a scale from 1 to 5] — Assessed with the Perceived Benefit sub-scale of the BSASabb (an abridged version of the Booster Seat Attitudes Scale, Cunningham et al., 2011). The Perceived Benefit subscale evaluates parents' perception of the general safety afforded by booster seats (e.g., prevents children from being injured during normal driving), on a scale from 1 to 5, where higher scores indicate the parent perceives more safety benefit afforded by booster seats.
  Scores on a scale from 1 to 5 | 4.31 (0.69) | 4.31 (0.70) | 4.31 (0.69)
Perceived key benefit of booster seats [Mean (Standard Deviation); unit: Scores on a scale from 1 to 5] — Assessed with the Key Benefit sub-scale of the BSASabb (an abridged version of the Booster Seat Attitudes Scale, Cunningham et al., 2011). The Key Benefit sub-scale evaluates parents' perception of the safety afforded by booster seats in relation to potentially fatal injuries to the spine and neck (a key feature of booster seats), on a scale from 1 to 5, where higher scores indicate the parent perceives more benefit afforded by booster seats..
  Scores on a scale from 1 to 5 | 4.45 (0.68) | 4.45 (0.64) | 4.45 (0.66)
Intent to use booster seats [Mean (Standard Deviation); unit: Scores on a scale from 1 to 5] — Assessed with the Intent to Use sub-scale of the BSASabb (an abridged version of the Booster Seat Attitudes Scale, Cunningham et al., 2011). Intent to Use sub-scale evaluates parents' willingness to purchase and ensuring their child always rides on a booster seat, on a scale from 1 to 5, where higher scores indicate the parent has more willingness to ensure their child always rides on a booster seat.
  Scores on a scale from 1 to 5 | 4.73 (0.50) | 4.69 (0.52) | 4.71 (0.51)
Intent to Learn about booster seats [Mean (Standard Deviation); unit: Scores on a scale from 1 to 5] — Assessed with the Intent to Learn sub-scale of the BSASabb (an abridged version of the Booster Seat Attitudes Scale, Cunningham et al., 2011). Intent to Learn sub-scale evaluates parents' willingness to attend to a booster seat clinic or workshop, on a scale from 1 to 5, where higher scores indicate the parent has more willingness to attend clinics or workshops on booster seats.
  Scores on a scale from 1 to 5 | 3.63 (1.09) | 3.65 (1.02) | 3.64 (1.05)

OUTCOME MEASURES:

1. Primary Outcome: Change in Perceived Safety Benefit of Booster Seats
Description: Assessed with the Perceived Benefit sub-scale of the BSASabb (an abridged version of the Booster Seat Attitudes Scale, Cunningham et al., 2011). The Perceived Benefit subscale evaluates parents' perception of the general safety afforded by booster seats (e.g., prevents children from being injured during normal driving). The Perceived Benefit sub-scale of the BSASabb ranges from 1 to 5, and higher scores mean better outcome.
Time Frame: Immediately before intervention; immediately after intervention (the mean duration of the intervention was 3 minutes)
Population: Only participants with complete data in the Perceived Benefit sub-scale of the BSASabb were included.
Measure: Mean (Standard Deviation); unit: Scores on a scale from 1 to 5
Arm/Group | Current Material | Enhanced Material
Number analyzed (Participants) | 360 | 357
Scores on a scale from 1 to 5 | 0.27 (0.53) | 0.15 (0.53)
Statistical Analysis 1: Comparison: Current Material vs Enhanced Material; Test type: Superiority; p = 0.002, t-test, 2 sided — Threshold for significance: <0.05; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [0.04 to 0.20]

2. Primary Outcome: Change in Key Benefit of Booster Seats
Description: Change in key safety was measured as the difference between post- and pre-intervention scores assessed with the Key Benefit sub-scale of the BSASabb (an abridged version of the Booster Seat Attitudes Scale, Cunningham et al., 2011). The Key Benefit sub-scale evaluates parents' perception of the safety afforded by booster seats in relation to potentially fatal injuries to the spine and neck, a key feature of booster seats. The Key Benefit sub-scale of the BSASabb ranges from 1 to 5 and higher scores mean better outcome.
Time Frame: Immediately before intervention; immediately after intervention (the mean duration of the intervention was 3 minutes)
Population: Only participants with complete data in Key Benefit sub-scale of the BSASabb were included.
Measure: Mean (Standard Deviation); unit: Scores on a scale from 1 to 5
Arm/Group | Current Material | Enhanced Material
Number analyzed (Participants) | 360 | 356
Scores on a scale from 1 to 5 | 0.29 (0.54) | 0.15 (0.50)
Statistical Analysis 1: Comparison: Current Material vs Enhanced Material; Test type: Superiority; p = 0.000, t-test, 2 sided — Threshold for significance: 0.05; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [0.07 to 0.22]

3. Secondary Outcome: Change in Intention to Use Booster Seats
Description: Change in intention to use booster seats was measured as the difference between post- and pre-intervention scores in the Intent to Use sub-scale of the BSASabb (an abridged version of the Booster Seat Attitudes Scale, Cunningham et al., 2011). Intent to Use sub-scale evaluates parents' willingness to purchase and ensuring their child always rides on a booster seat. The Intention to Use of the BSASabb ranges from 1 to 5 and higher scores mean better outcome.
Time Frame: Immediately before intervention; immediately after intervention (the mean duration of the intervention was 3 minutes)
Population: Only participants with complete data in the Intent to Use sub-scale of the BSASabb were included.
Measure: Mean (Standard Deviation); unit: Scores on a scale from 1 to 5
Arm/Group | Current Material | Enhanced Material
Number analyzed (Participants) | 360 | 360
Scores on a scale from 1 to 5 | 0.03 (0.38) | 0.01 (0.32)
Statistical Analysis 1: Comparison: Current Material vs Enhanced Material; Test type: Superiority; p = 0.352, t-test, 2 sided — Threshold for significance: 0.05; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.03 to 0.07]

4. Secondary Outcome: General Knowledge of Booster Seats
Description: Participants were asked questions to assess how much general information about booster seats they retained: how booster seats prevent injuries as well as guidelines and recommendations. Scores ranges from 0 to 2 and higher scores mean better outcome.
Time Frame: immediately after intervention (the mean duration of the intervention was 3 minutes)
Population: Only participants with complete data on general knowledge of booster seats were included.
Measure: Mean (Standard Deviation); unit: score on a scale from 0 to 2
Arm/Group | Current Material | Enhanced Material
Number analyzed (Participants) | 360 | 352
score on a scale from 0 to 2 | 0.83 (0.70) | 1.29 (0.74)
Statistical Analysis 1: Comparison: Current Material vs Enhanced Material; Test type: Superiority; p = 0.000, t-test, 2 sided — Threshold for significance: <0.05; Mean Difference (Final Values) = 0.45, 95% CI 2-sided [0.34 to 0.56]

5. Secondary Outcome: Projected Intent to Use
Description: Participants were asked to estimate how likely were their peers to use about booster seats, after reviewing the information they were assigned. The questionnaire was based on the Booster Seat Attitudes Scale (Cunningham et al., 2011). The idea behind this measure is that people judgments about what others would do reflect, in part, what they would do (Loewenstein, 2005). The scale ranges from 1 to 5 and higher scores mean better outcome.
Time Frame: Immediately after intervention (the mean duration of the intervention was 3 minutes)
Population: Only participants with complete data on the Projected Intent to use scale were included in this analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale from 1 to 5
Arm/Group | Current Material | Enhanced Material
Number analyzed (Participants) | 360 | 360
Scores on a scale from 1 to 5 | 4.46 (0.62) | 4.62 (0.53)
Statistical Analysis 1: Comparison: Current Material vs Enhanced Material; Test type: Superiority; p = 0.002, t-test, 2 sided — Threshold for significance: 0.05; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [0.05 to 0.22]

6. Secondary Outcome: Interest in the Communication Material
Description: Number of seconds spent reviewing the material.
Time Frame: Immediately after intervention (the mean duration of the intervention was 3 minutes)
Population: Only participants who completed their assigned material were included in this analysis.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Current Material | Enhanced Material
Number analyzed (Participants) | 360 | 360
Seconds | 161 (190) | 128 (218)
Statistical Analysis 1: Comparison: Current Material vs Enhanced Material; Test type: Superiority; p = 0.033, t-test, 2 sided — Threshold for significance: <0.05; Mean Difference (Final Values) = 32.56, 95% CI 2-sided [2.65 to 62.46]

7. Secondary Outcome: Interest in Additional Information
Description: Whether parents review additional information offered as external links to legislation, car seat clinics, and list of product recalls. Measured as "Yes" or "No".
Time Frame: Immediately after intervention (the mean duration of the intervention was 3 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Current Material | Enhanced Material
Number analyzed (Participants) | 364 | 367
Participants
  Clicked links to additional information on booster seats | 17 | 26
  Did not clicked links to additional information on booster seats | 347 | 341

8. Secondary Outcome: Applied Knowledge of Booster Seats
Description: Participants were shown a picture of a child incorrectly restrained and were asked to identify the mistakes in the picture. Scores ranges from 0 to 3 and higher scores mean better outcome.
Time Frame: Immediately after intervention (the mean duration of the intervention was 3 minutes)
Population: Only participants with complete data on general knowledge of booster seats were included.
Measure: Mean (Standard Deviation); unit: score on a scale from 0 to 3
Arm/Group | Current Material | Enhanced Material
Number analyzed (Participants) | 359 | 360
score on a scale from 0 to 3 | 2.60 (0.68) | 2.70 (0.64)
Statistical Analysis 1: Comparison: Current Material vs Enhanced Material; Test type: Superiority; p = 0.065, t-test, 2 sided — Threshold for significance: <0.05; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [0.00 to 0.19]

9. Secondary Outcome: Projected Intent to Learn
Description: Participants were asked to estimate how likely were their peers to learn about booster seats, after reviewing the information they were assigned. The questionnaire was based on the Booster Seat Attitudes Scale (Cunningham et al., 2011). The idea behind this measure is that people judgments about what others would do reflect, in part, what they would do (Loewenstein, 2005). The scale ranges from 1 to 5 and higher scores mean better outcome.
Time Frame: Immediately after intervention (the mean duration of the intervention was 3 minutes)
Population: Only participants with complete data on the Projected Intent to Learn scale were included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale from 1 to 5
Arm/Group | Current Material | Enhanced Material
Number analyzed (Participants) | 360 | 360
units on a scale from 1 to 5 | 3.81 (0.91) | 3.95 (0.89)
Statistical Analysis 1: Comparison: Current Material vs Enhanced Material; Test type: Superiority; p = 0.030, t-test, 2 sided — Threshold for significance: <0.05; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [0.01 to 0.28]

ADVERSE EVENTS:
Time Frame: Since this is an educational intervention, data on adverse events (as defined by ClinicalTrials.gov) were not collected.
Description: Since this is an educational intervention, data on adverse events (as defined by ClinicalTrials.gov) were not collected. We collected information of whether participants misunderstood the information the information provided does not fall under any of the categories specified by ClinicalTrials.gov (Misunderstanding of information cannot be grouped by organ system, for example).
Groups:
- All Participants: All participants who reviewed education material as part of their assigned intervention, regardless of their alocation.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
First: It is difficult to determine if findings are behaviorally meaningful, because the instruments used are new. Second: The presence of ceiling effects indicate that the effect was underestimated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-06-27): https://cdn.clinicaltrials.gov/large-docs/30/NCT03573830/Prot_SAP_ICF_000.pdf